CLINICAL TRIAL: NCT01079091
Title: Hepa Wash Treatment of Patients With Acute-on-Chronic Liver Failure in Intensive Care Units
Acronym: HEPATICUS-1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The foundations of our pilotstudy planning has changed.
Sponsor: Hepa Wash GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS001
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Acute on Chronic Hepatic Failure
Keywords: Liver failure; Hepatic insufficiency; Liver Cirrhosis; Artificial liver; Albumin dialysis
MeSH Terms: conditions — Liver Failure; Hepatic Insufficiency; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADVOS (Hepa Wash) (Experimental): Treatment with the liver support system "Hepa Wash"
  Interventions: Device: ADVOS (Hepa Wash); Procedure: Standard Medical Therapy

INTERVENTIONS:
Device: ADVOS (Hepa Wash) — Intervention frequency: 1-10 treatments (decision of the investigator)
  Duration of intervention per patient: Treatment until recovery or death (max. 6 weeks)
  Other Names: Hepa Wash procedure; the HIP1001 system
Procedure: Standard Medical Therapy — Standard of care treatment

SUMMARY:
Patients with compensated chronic liver disease who have an episode of acute deterioration of liver function (acute-on-chronic liver failure) are known to have up to 90% mortality rate. Hepa Wash(R) is a newly developed liver and renal support system that is based on the use of recycled albumin dialysate. The new system has shown a high detoxification capacity in in-vitro and preclinical studies. The aim of the study is to evaluate the safety and efficacy of the Hepa Wash system in patients with acute-on-chronic liver failure in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented clinical or histological evidence of cirrhosis AND
2. Acute decompensation in previously stable cirrhotic liver disease AND
3. Bilirubin ≥ 2 mg/dl AND
4. SOFA ≥ 9 calculated after 12 hours of optimal medical therapy AND
5. Patient is in the intensive care unit AND
6. Informed consent of the patient or the legal representative AND
7. Patients are 18y or older AND
8. Enrollment of patients within 96 hours of fulfilling inclusion criteria (1-5)

Exclusion Criteria:

1. Untreatable extrahepatic cholestasis
2. Patient has a survival prognosis of less than 6 weeks because of a chronic disease (e.g. metastasizing cancer) and before the acute event which lead to the ICU admission.
3. PaO2/FIO2 ≤ 100 mmHg (respiratory SOFA-score of 4)
4. Patients who receive a vasopressor support of Dopamine >15 µg/kg/min or epinephrine >0.1 µg/kg/min or norepinephrine >0.1 µg/kg/min (cardiovascular SOFA-score of 4)
5. Patients with creatinine ≥5 mg/dl or urine output <200 ml/day (renal SOFA-score of 4)
6. Patients on kidney dialysis
7. Patient with MELD-score of 40
8. Mean arterial pressure ≤ 50 mmHg despite conventional medical treatment
9. Patient testament excludes the use of life-prolonging measures
10. Post-operative patients whose liver failure is related to liver surgery
11. Uncontrolled seizures
12. Active or uncontrolled bleeding
13. Weight ≥ 120 kg
14. Pregnancy
15. Patient diagnosed with Creutzfeldt-Jakob disease
16. Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
30-day mortality rate | 30 days
  Mortality 30 days after the first intervention

SECONDARY OUTCOMES:
Multiorgan system failure according to Sequential Organ Failure Assessment (SOFA) Score | 72 hours
  The Sequential Organ Failure Assessment (SOFA) Score analyses the severity of illness according to 6 organ systems (CNS, Liver, Kidney, Hemodynamic, Coagulation, Lung). Each system is given 0 to 4 points for a total of 24 points. A value >2 in each of the systems indicates organ failure. An overall value > 14 indicates 90% probability of in-hospital mortality.
Safety (adverse events and surrogate parameters) | 30 days
  Adverse Events during the intervention will be assessed. Additionally, liver parameters (e.g. Bilirubin), Kidney Parameters (e.g. Creatinin, Urea) and blood gas analysis will be performed.
Number of days on ventilation | 30 days
  Number of days with need of mechanical ventilation after first intervention
Number of days without extracorporeal treatment | 30 days
  Number of days without the need of extracorporeal renal and/or liver replacement therapy after the first intervention
180d-mortality rate | 180 days
  Mortality 180 days after the first intervention
1y-mortality rate | 1 year
  Mortality 1 year after the first intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Huber, PD Dr., Principal Investigator — II Medizinische Klinik, Klinikum rechts der Isar, Munich
Locations (1):
- II Medizinische Klinik, Klinikum rechts der Isar, Munich, Bavaria, Germany

REFERENCES:
- [Result] Huber W, Henschel B, Schmid R, Al-Chalabi A. First clinical experience in 14 patients treated with ADVOS: a study on feasibility, safety and efficacy of a new type of albumin dialysis. BMC Gastroenterol. 2017 Feb 16;17(1):32. doi: 10.1186/s12876-017-0569-x. PMID 28209134